CLINICAL TRIAL: NCT05880537
Title: Safety, Efficacy, & Use of Decellularized Femoral Artery Allograft for Arteriovenous Access for Hemodialysis: A Multi-center Prospective Registry Study
Brief Title: Decellularized Femoral Artery Allograft (Nexeon AVX) Prospective Registry
Status: Recruiting | Type: Observational
Sponsor: LifeNet Health (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-21-005
Record Dates: First submitted 2023-03-01; First posted 2023-05-30 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Open Label: Open Label for subjects with End-Stage Renal Disease
  Interventions: Other: Nexeon Arterial Venous Allograft

INTERVENTIONS:
Other: Nexeon Arterial Venous Allograft — Nexeon AVX allograft for hemodialysis access in end stage renal disease

SUMMARY:
Post market registry to assess the safety and efficacy of a novel decellularized human femoral artery allograft (Nexeon AVX Decellularized Femoral Artery,

DETAILED DESCRIPTION:
The clinical objective of this prospective, observational, post market registry study, CR-21-005, is to assess the safety and efficacy of a decellularized human femoral artery allograft (Nexeon AVX Decellularized Femoral Artery, LifeNet Health, Virginia Beach, VA) in the creation of vascular access for hemodialysis in patients with ESRD.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female, ≥18 years of age at the time of graft placement
2. Have a diagnosis of ESRD or renal dysfunction requiring hemodialysis
3. Subject requires dialysis access to start or maintain dialysis treatment and placement of an AV access graft is a viable access option.
4. Have the ability themselves, or through their legal guardian, to understand the requirements of the study, to provide written informed consent/assent as evidenced by signature on an informed consent form (ICF) approved by an institutional review board (IRB), and to agree to abide by the study restrictions and return to the site for the required assessments
5. Have provided written authorization for use and disclosure of protected health information

Exclusion Criteria:

1. Be participating in a study of another investigational drug or device
2. Have a known sensitivity to any of the processing reagents utilized in the manufacture of this product such as antibiotics (Lincomycin, Polymyxin B, Ciprofloxacin, Meropenum, Gentamicin, or Vancomycin) and processing reagents (N-lauroyl sarcosine, Denarase and glycerol/glycerin)
3. Have a history or evidence of severe cardiac disease, myocardial infarction within 6 months, ventricular arrhythmias, or unstable angina requiring continuing treatment
4. Have a history or evidence of severe peripheral vascular disease in the upper extremities
5. Have the inability or be unable or unwilling to follow the study visit schedule
6. Have the presence of any condition that, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry subject population will consist of male and female research subjects, 18 years of age or older at the time of graft placement, who require vascular access for hemodialysis that the surgeon determines, in their medical judgement, to be a candidate to receive the Nexeon AVX graft. The target study enrollment is 100 subjects. Each subject will be followed for a maximum of two (2) years or 24 months post-graft placement.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
UltraSound evaluation of allograft functional patency. | 24 months
  Ultrasound proof of vessel patency and blood flow

SECONDARY OUTCOMES:
Secondary Endpoint: | 24 months
  Evaluating the emergent adverse events as it pertains to the hemodialysis access anatomical site

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Infirmary Heath, Mobile, Alabama
  - Olive View - UCLA Medical Center, Sylmar, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Sentara Norfolk General Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No